CLINICAL TRIAL: NCT03928795
Title: Perinatal Morbidity Factors During Elective Cesarean Section
Brief Title: Perinatal Morbidity Factors During Cesarean Section
Status: Completed | Type: Observational
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Kaouther Dimassi, associate professor in obstetrics and gynecoloy, University Tunis El Manar
Other Study IDs: perinatal morbidity mongi slim
Record Dates: First submitted 2019-04-23; First posted 2019-04-26 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Perinatal Morbidity
Keywords: neonatal ph; neonatal eucapnic ph; fetal extraction; elective caesarean; apgar score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- neonates with acute acidosis: neonates with Cord blood gases measured immediately after birth inferior to 7.15
  Interventions: Procedure: elective caesarean section
- neonates with a normal ph: neonates with Cord blood gases measured immediately after birth of at least 7.15
  Interventions: Procedure: elective caesarean section

INTERVENTIONS:
Procedure: elective caesarean section — elective caesarean section

SUMMARY:
Caesarean section is one of the most common surgeries in the world and the increasing rate of cesarean delivery is associated with increased maternal and fetal morbidity when compared to vaginal delivery.

With this dramatic increase in caesarean section rates, it is urgent to identify factors that may affect perinatal morbidity. Indeed, such factors can be classified into:

* Modifiable factors: surgical technique, anesthesia technique, operator experience, operative time
* Not modifiable factors: characteristics inherent to the mother: BMI, gravidic pathology, number of caesareans...

Majority of previous studies focused on anesthetic factors. A global vision integrating all parameters is necessary in order to best guide the preventative measures to be put in place.

our Objectives were : To Identify and to Analyze Perinatal Morbidity Factors During Caesarean Section

DETAILED DESCRIPTION:
I- Characteristics of the study:

Non-interventional descriptive longitudinal prospective study.

II- Location and period of study:

The study tooked place in the obstetrics and gynecology department of the Mongi Slim La Marsa University Hospital from 27 august 2018 until 10.04.2019.

III- The study population:

Was defined by all women with indication of an elective caesarean section in our department during the study period.

IV-The eligibility criteria:

1. The inclusion criteria:

   * Monofetal pregnancy
   * Age over 18 years old
   * Term Pregnancy ≥ 37SA
   * Elective caesarean section
2. The non-inclusion criteria:

   * Fetal pathology known prenatally like intrauterine severe growth retardation with Doppler abnormalities, fetal malformation or a known fetal genetic defect.
   * Anomaly of placental adhesion.
   * Caesarean in a context of medical or obstetric emergency.
3. Exclusion criteria:

   * Caesarean section performed under general anesthesia following failure of locoregional anesthesia.
   * Refusal of the woman to participate in the study.
   * Impossibility or failure to study the neonatal acid-base balance on the umbilical cord.

V-Investigators:

1. The resident responsible for the study :

   He was responsible for the inclusion and collection of preoperative and postoperative data.
2. Surgeons :

They immediately after surgery reported on the patient information sheet the surgical features of the cesarean section: the technique used, the methods of fetal extraction, the difficulties encountered...

VI- The judgment criteria:

* The acid-base balance of the newborn that will be evaluated by the measurement of neonatal PH at the umbilical cord and the neonatal eucapnic [1-2-3].
* The APGAR score at 5 minutes [4]
* Rates of transfer to neonatal intensive care unit ( NICU) and reason for hospitalization.

VII-The progress of the study:

1. The pre-inclusion visit

   All the patients followed at the outpatient clinic were informed of the study during the prenatal visit of the 8th month.

   The resident responsible for the study checked the eligibility criteria and informed the patient of the research objectives, its progress and the expected benefits of the research.

   He answered all questions about Cesarean the study. A period of reflection until the day of delivery was left for signing the consent form. (see annexes 1 and 2)
2. The inclusion visit The resident in charge of the study was responsible for the final verification of the eligibility criteria and obtaining the written informed consent of the patient in Arabic (Appendix 1) and in French (Appendix 2).

   If the patient agreed to participate, the investigator wrote his name and surname in clear, date and sign the consent form.

   The patients recruited were chronologically assigned a number until the end of the study.
3. The day of cesarean section Once the patient had been selected for the study, her delivery was planned according to gestational age and respected the usual recommendations and protocols of use in the department.

Thus, the indication of cesarean delivery and the date of the operation were not affected by the inclusion of the patient in this observational study.

Investigators described the anesthetic and surgical techniques. Thus, the patient file was completed prospectively and specified the items relating to

* The surgeon:

The rank of the operator and his experience in caesarean surgery.

-Caesarean technique: Indeed, two caesarean techniques are used in our department and the choice between the two was attributed to the operator.

* The intraperitoneal Misgav Ladach technique [5]
* Extraperitoneal caesarean section according to the technique "French ambulatory cesarean section" (FAUCS) [6]
* The different operating times:
* Time between the beginning of the anesthesia and the incision of the skin.
* Time between skin incision and fetal extraction.
* Time between hysterotomy and fetal extraction or actual duration of fetal extraction.
* The modalities of fetal extraction:
* fetal presentation
* Possible use of instruments
* Use of maneuvers for intraoperative fetal extraction
* Operator's subjective evaluation of the degree of difficulty encountered to achieve fetal extraction
* Neonatal outcome:
* The neonatal PH measured at the umbilical cord.
* The eucapnic neonatal PH.
* The Apgar score at 5 minutes.
* Possible hospitalization in neonatology department and in which case its reason.

VIII-Statistic study:

We performed a correlation Pearson study between the different operating times measured during the study and the value of the neonatal eucapnic PH.

We performed a logistic regression to identify among the used variables the factors that significantly and independently influenced the neonatal outcome. We identified two major events : neonatal ph<7.15 and neonatal ph <7.1

ELIGIBILITY:
Inclusion Criteria:

* Monofetal pregnancy
* Age over 18 years old
* Term Pregnancy ≥ 37SA
* Indication for Elective caesarean section

Exclusion Criteria:

* -Fetal pathology known prenatally like intrauterine severe growth retardation with Doppler abnormalities, fetal malformation or a known fetal genetic defect.
* Anomaly of placental adhesion.
* Caesarean in a context of medical or obstetric emergency.
* Caesarean section performed under general anesthesia following failure of locoregional anesthesia.
* Refusal of the woman to participate in the study.
* Impossibility or failure to study the neonatal acid-base balance on the umbilical cord.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Was defined by all women with indication of an elective caesarean section in our department during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
neonatal acid base balance | immediately after fetal extraction
  Cord blood gases

SECONDARY OUTCOMES:
apgar score | 1,3,5 and 10 minutes of life
  The Apgar score is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. The five criteria are summarized using words chosen to form an ackronym (Appearance, Pulse, Grimace, Activity, Respiration).he test is generally done at 1 and 5 minutes after birth and may be repeated later if the score is and remains low. Scores 7 and above are generally normal; 4 to 6, fairly low; and 3 and below are generally regarded as critically low and cause for immediate resuscitative efforts.

OTHER OUTCOMES:
neonatal transfer to neonatal intensive care unit | during the first day
  hospitalisation in intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: kaouther simassi, MD, Principal Investigator — university tunis el manar , faculty of medicine Tunis, TUNISIA
Locations (1):
- Kaouther Dimassi, Tunis, Sidi Daoued La Marsa, Tunisia